CLINICAL TRIAL: NCT06648239
Title: Coronary Computed Tomographic Angiography to Optimize Diagnostic Yield of Invasive Angiography for Low-risk Patients Screened With Artificial Intelligence
Brief Title: CCTA to Optimize Diagnostic Yield of Invasive Angiography With AI
Acronym: CarDIA-AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 17103
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: Artificial Intelligence (AI); Coronary Angiography; Coronary Computed Tomography Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will proceed directly to ICA as originally referred.
  Interventions: Other: Usual Care
- Centralized triage with risk score-based screening for obstructive CAD (Experimental): Patients originally referred for ICA will be screened for obstructive CAD with a decision support tool that uses data from their referral forms. Patients will receive either CCTA or ICA based on their predicted probability of obstructive CAD.
  Interventions: Other: Centralized triage with risk score-based screening for obstructive CAD

INTERVENTIONS:
Other: Usual Care — In the usual care group, patients will proceed directly to ICA following referral from community cardiology, as is the current standard of care. Research staff will screen participants in this group for significant CAD using the decision support tool; however, the tool's recommendations will not affect their care, as all patients in this group will invariably receive ICA.
  Arms: Usual Care
Other: Centralized triage with risk score-based screening for obstructive CAD — Patients randomized to the intervention will have selected features of their medical history, recorded on their referral form, entered into a decision support tool by research personnel to generate a recommendation of whether they should proceed directly to ICA or whether they should receive CCTA. Patients with recommendations for ICA will proceed directly to ICA. Patients with recommendations for CCTA will be referred to CCTA. Based on the results of the CCTA, recommendations for medical management versus referral for ICA will be made.
  Arms: Centralized triage with risk score-based screening for obstructive CAD

SUMMARY:
Coronary artery disease (CAD) is a leading cause of death. The gold-standard test used to diagnose CAD is invasive coronary angiography (ICA). However, nearly half the patients who receive ICA are found to have no disease or non-significant disease. This means that while they receive a diagnosis, they do not receive any therapeutic benefit. This is concerning because ICA is expensive and it carries a risk to patients. A non-invasive diagnostic test, cardiac computed tomographic angiography (CCTA), has been shown to be as effective as ICA at diagnosing CAD in the right patient population, while being less expensive and less risky for patients. An optimal solution would involve screening to identify which patients are good candidates for CCTA vs. which should receive ICA. This screening tool could be used in a triage pathway to ensure that every patient gets the test that is best for them. The investigators have used Artificial Intelligence (AI) to develop a model for determining which patients should receive ICA vs. which should receive CCTA. The investigators have also developed a triage pathway to direct patients to the most appropriate test. The investigators now plan to evaluate the AI tool combined with the triage pathway through a clinical trial at Hamilton Health Sciences and Niagara Health. This model of care will reduce risk to patients, reduce wait times for ICA and reduce costs to the health care system.

ELIGIBILITY:
Inclusion Criteria

Patients are eligible if they:

1. are ≥18 years of age;
2. are referred for non-urgent (elective) outpatient ICA;
3. have an indication for ICA that includes 'Rule out CAD', 'Cardiomyopathy', or 'Stable CAD'; and
4. are able to provide informed consent in English.

Exclusion Criteria Patients are ineligible if they have:

1. received a prior high-quality coronary computed tomographic angiography (CCTA) within the last 5 years;
2. atrial fibrillation;
3. known severe renal dysfunction (GFR <35);
4. planned non-coronary cardiac surgery;
5. any prior obstructive CAD, acute coronary syndrome, percutaneous coronary intervention, or coronary artery bypass graft; or
6. known severe coronary artery calcification (calcium score >1000).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of normal/non-obstructive CAD diagnosed through ICA | 90 days (after randomization)
  The rate of normal or non-obstructive CAD diagnosed through ICA in patients referred for cardiac investigation. The rate for an arm (control vs experimental) is calculated by dividing the number of patients diagnosed with normal/non-obstructive CAD through ICA by the total patients allocated to the arm.

SECONDARY OUTCOMES:
Quantitative assessment of number of angiograms avoided | 90 days (after randomization)
  Number of angiograms avoided due to CCTA bookings.
Deviation from management recommendations following CCTA (i.e. angiograms performed when not recommended) | 90 days (after randomization)
  Number of angiograms performed when not recommended.
Diagnostic yield of invasive angiography | 90 days (after randomization)
  Diagnostic yield is defined as the proportion of invasive angiograms that identify significant disease (≥70% stenosis) on a major coronary vessel (>2 mm) or >50% stenosis in the left main).
Sex differences in rate of normal/non-obstructive CAD diagnosed through ICA | 90 days (after randomization)
  Difference in the rate of normal/non-obstructive CAD diagnosed through ICA between males and females.
Site differences in rate of normal/non-obstructive CAD diagnosed through ICA | 90 days (after randomization)
  Difference in the rate of normal/non-obstructive CAD diagnosed through ICA between sites.
Budget impact of new strategy for risk stratification of CAD in low-risk patients | 90 days (after randomization)
  Cost of risk stratification of CAD in low risk patients.
Number of low-quality CCTAs | 90 days (after randomization)
  The quality will be graded on a per-patient basis using a three-class system: low quality, denoting an image in which the coronary anatomy cannot be clearly defined, requiring ICA within 90 days for clarification; suboptimal quality, denoting an image in which the coronary anatomy was equivocal for one or more non-prognostic vessels but not requiring ICA based on CCTA findings and clinical presentation; and high quality, denoting an image in which the coronary anatomy could be clearly defined.

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David Schwalm, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation; Jeremy Petch, PhD, Principal Investigator — Hamilton Health Sciences Corporation; Natalia Pinilla-Echeverri, MD, PhD, Principal Investigator — Niagara Health
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Catharines Hospital, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwalm JD, Di S, Sheth T, Natarajan MK, O'Brien E, McCready T, Petch J. A machine learning-based clinical decision support algorithm for reducing unnecessary coronary angiograms. Cardiovasc Digit Health J. 2021 Dec 24;3(1):21-30. doi: 10.1016/j.cvdhj.2021.12.001. eCollection 2022 Feb. PMID 35265932
- [Background] Schwalm JD, Bouck Z, Natarajan MK, Pinilla N, Walker D, Syed N, Landry D, Sabri A, Tandon V, Nkurunziza J, Taljaard M, Sheth T. Centralized Triage of Suspected Coronary Artery Disease Using Coronary Computed Tomographic Angiography to Optimize the Diagnostic Yield of Invasive Angiography. CJC Open. 2022 Nov 19;5(2):148-157. doi: 10.1016/j.cjco.2022.10.009. eCollection 2023 Feb. PMID 36880068
- [Background] Schwalm JD, Sheth T, Pinilla-Echeverri N, Petch J. Using Artificial Intelligence to Optimize the Use of Cardiac Investigations in Patients With Suspected Coronary Artery Disease. J Soc Cardiovasc Angiogr Interv. 2024 Mar 26;3(3Part B):101305. doi: 10.1016/j.jscai.2024.101305. eCollection 2024 Mar. No abstract available. PMID 39131228
- [Derived] Petch J, Tabja Bortesi JP, Sheth T, Natarajan M, Pinilla-Echeverri N, Di S, Bangdiwala SI, Mosleh K, Ibrahim O, Bainey KR, Dobranowski J, Becerra MP, Sonier K, Schwalm JD. Coronary Computed Tomographic Angiography to Optimize the Diagnostic Yield of Invasive Angiography for Low-Risk Patients Screened With Artificial Intelligence: Protocol for the CarDIA-AI Randomized Controlled Trial. JMIR Res Protoc. 2025 May 21;14:e71726. doi: 10.2196/71726. PMID 40397500